# A Critical Analysis of Anaplastic Thyroid Clinical Trials: Perspectives from Patient Experiences

Informed Consent Form (ICF) For <u>Power Clinical Trial's</u> Anaplastic Thyroid Trial

Date: April 6, 2023

An Overview of the Informed Consent Form

The informed consent form (ICF) is an essential document that plays a critical role in the clinical trial process. It is designed to ensure that potential participants are fully informed about the study they are considering participating in, and that they provide voluntary consent to take part in the research. The ICF is divided into two distinct parts, each serving a specific purpose.

The first part of the ICF is the Patient Information Sheet, which contains detailed information about the clinical study. This section covers key aspects of the study, including its purpose, design, procedures, potential risks and benefits, and your role as a participant. It is essential that you take the time to read and understand this section thoroughly, as it will enable you to make an informed decision about whether to participate in the study or not.

The second part of the ICF is the Certificate of Consent, which serves as written evidence of your agreement to participate in the study. By signing the Certificate of Consent, you are indicating that you have read and understood the Patient Information Sheet and that you agree to participate in the study voluntarily.

It is important to note that your signature does not waive your legal rights or commit you to continue participation in the study. You are free to withdraw from the study at any time, without any negative consequences.

Once you have completed the ICF and signed the Certificate of Consent, you will receive a copy of the document for your records. This copy will serve as a reminder of

the information provided, and of your decision to participate in the study. It is important that you keep this copy safe, as you may need to refer back to it at a later stage.

## Overview of the Anaplastic Thyroid Cancer Clinical Trial

Anaplastic thyroid cancer is an uncommon and dangerous kind of thyroid cancer that develops from the thyroid gland's follicular cells. Even though it only represents 2% of thyroid cancer cases, it is the main cause of thyroid cancer-related fatalities. Treatment options for anaplastic thyroid carcinoma are few and difficult to administer. Clinical trials, however, give promise for the creation of novel and enhanced therapies that can enhance patient outcomes and quality of life.

Clinical studies for anaplastic thyroid carcinoma are crucial, and this cannot be stressed enough.

These trials allow researchers to explore novel therapeutics that might not be accessible through conventional treatment choices and provide them crucial insights into the underlying causes of the disease. Also, clinical trials provide patients the chance to obtain advanced medical care from top medical specialists and access cutting-edge medicines.

Ensuring that clinical trial participation percentages appropriately reflect the greater community of patients with anaplastic thyroid carcinoma is crucial. Sadly, underrepresented groups may have lower participation rates as a result of a variety of issues, including limited information availability, mistrust of the healthcare system, and communication difficulties. This clinical study intends to comprehend these variables and find methods to boost trial participation rates in the future.

Our goal is to raise clinical trial participation rates by determining and comprehending the causes of underrepresented groups' low participation rates. We think that by identifying these variables, we can create more effective plans for raising participation rates in upcoming clinical trials.

It is crucial to understand that taking part in this clinical experiment is completely voluntary, and participants are free to leave at any moment without facing any repercussions. The participants face little danger throughout the study's principal procedures, which include responding to surveys and placing follow-up calls. Before choosing, we advise prospective participants to thoroughly read the permission form and consult with their loved ones, close friends, trusted advisers, and medical

specialists. You may further your understanding of anaplastic thyroid carcinoma by taking part in this study.

## The Research Methodology

This clinical trial is designed as an observational study and does not involve any changes to your current treatment plan. If you choose to participate, the researcher will conduct interviews to collect data, but they cannot diagnose or recommend any treatment. The study's goal is to gather information to improve understanding of the disease and help develop better treatments in the future.

#### **Enrolment in the Clinical Trial**

This study requires you to be currently enrolled in another clinical trial for anaplastic thyroid cancer to participate. Our aim is to gain a better understanding of why patients choose to take part in this type of research and what factors affect their decision to continue or stop treatment.

We are interested in learning about the factors that led you to participate in the study and what influences your decision to continue or discontinue. The goal of this clinical trial is to identify the factors that influence patient decision-making in anaplastic thyroid cancer clinical trials.

Participation in this study is voluntary and optional, and will not impact your current treatment plan in another clinical trial. If you feel uncomfortable or wish to withdraw from the study, you are free to do so at any time without any effect on your legal rights.

# Comparison to Other Anaplastic Thyroid Cancer Clinical Trials

There are many interventional clinical trials available for patients with anaplastic thyroid cancer, but this particular trial is different. Rather than requiring participation in a specific treatment plan, this trial is purely observational in nature.

It's important to note that there is numerous other research available, and while we cannot list them all here, interested individuals can visit clinicaltrials.gov for a

comprehensive list of <u>anaplastic thyroid cancer studies</u> or Power's website to explore their options for <u>anaplastic thyroid cancer clinical trials</u>.

## What to Expect as a Participant

Should you choose to enroll in this clinical trial, you will be required to complete a survey every other week. Each survey usually takes around 30 minutes to complete. We will also have check-in calls with you every three months.

It is important to note that while you may need to be involved in another clinical trial that involves treatment, this particular study is strictly for observational purposes only. It will not impact your diagnosis or treatment plan for the other trial. If you have any questions about the other trial, please contact your personal healthcare team.

We respect your privacy, and you are not required to answer any questions that make you uncomfortable. You have the option to complete the survey on your own, or someone can read the questions to you and you can respond verbally. If you wish, you can skip any questions that you do not want to answer.

All of the information you provide will be kept completely anonymous. Your name will not be attached to the survey forms, and the data we collect will be confidential.

Please rest assured that any personal data you provide will be handled with the utmost care and kept strictly confidential. We will protect your privacy by using encryption, passwords, and anonymity measures, such as numerical identifiers instead of names, to ensure the anonymity of patients. Phone logs and digital permission forms will also be handled securely.

## Further Information on Diversity in Clinical Trials

To learn more about the topic of diversity and representation in clinical trials, we recommend reviewing the following published studies. They provide valuable insights and analysis on the importance of recruiting a diverse participant pool, as well as strategies for improving representation:

Gray, Darrell M., Timiya S. Nolan, John Gregory, and Joshua J. Joseph. "Diversity in clinical trials: an opportunity and imperative for community engagement." *The Lancet Gastroenterology & Hepatology* 6, no. 8 (2021): 605-607.

Woodcock, Janet, Richardae Araojo, Twyla Thompson, and Gary A. Puckrein. "Integrating research into community practice—toward increased diversity in clinical trials." New England Journal of Medicine 385, no. 15 (2021): 1351-1353.

### Patient's Statement

By signing below, I acknowledge that I have been selected to participate in an interventional clinical trial for patients with anaplastic thyroid cancer. I have carefully reviewed and fully understand the consent document, and any questions or concerns I may have had have been addressed to my satisfaction. I freely and voluntarily agree to take part in this study, and understand that my participation is entirely optional and that I may withdraw at any time without penalty.

I also acknowledge that my personal information will be kept confidential and that any data collected during the study will be kept secure.

| Participant's Signature | | |
|-------------------------|--------------------------|------|
| Name of Participant | Signature of Participant | Date |

## Statement of Person Responsible to Get Consent

It was my responsibility to obtain the participant's consent for their participation in the study, and I took the necessary measures to ensure that they understood all aspects of the study. This included explaining the details of the consent form in a clear and thorough manner and giving them ample time to ask any questions they may have had. I can confirm that the participant made their decision to participate in the study voluntarily and without any coercion or undue influence from me or anyone else. Finally, I provided the participant with a copy of the consent form for their reference.

| Signature of the Person | Responsible to Get Consent | t |
|-------------------------|----------------------------|----------|
| Name of Researcher | Signature of Researcher | <br>Date |